CLINICAL TRIAL: NCT03613571
Title: A Single-centre, Open Single-arm Study Where the Safety, Tolerability and Efficacy of Subcutaneously Administered ILB Will be Evaluated in Patients With Amyotrophic Lateral Sclerosis
Brief Title: A Study to Evaluate the Safety, Tolerability and Efficacy of ILB in Patients With Amyotrophic Lateral Sclerosis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Inclusion was stopped with 13 of 15 patients recruited according to protocol. Patients responded with no safety signals. Study stop was due to slow recruitment.
Sponsor: TikoMed AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1.5, 2019-06-25; 2017-005065-47 (EudraCT Number)
Record Dates: First submitted 2018-06-15; First posted 2018-08-03 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ILB (Experimental): ILB treatment
  Interventions: Drug: ILB

INTERVENTIONS:
Drug: ILB — The investigational medicinal product ILB will be given as single short-term s.c. injections in the abdomen, the thigh or the buttock, in that order of priority. Subjects will be observed for at least 3 hours after injection.The IMP is a sterile, colourless to pale yellow solution for subcutaneous injection.

SUMMARY:
This is a Phase 2a single-centre, open single-arm study in patients with Amyotrophic Lateral Sclerosis (ALS) of intermediate progression rate. Eligible subjects will be administered weekly doses of ILB. A total of 5 subcutaneous (s.c.) doses will be administered at the study clinic.

The study consists of 10 visits; One 2-part screening visit, 5 ILB administration visits, and 3 follow-up visits. Each individual patient's study participation will be 4 months, including the screening and follow-up visits. Fifteen patients are planned to be included.

The primary objective of the study is to evaluate the safety and tolerability of ILB in patients diagnosed with ALS.

ILB is a solution for subcutaneous (s.c.) injection in saline solution. The dose administered will depend on the subject's body weight at the second study visit, prior to the first ILB administration.

No formal sample size calculation has been performed for this study. The proposed sample size is considered sufficient in this early phase 2 development to provide adequate information on the patients. Categorical data will be presented as counts and percentages. Continuous data will be summarised using descriptive statistics.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to give written informed consent for participation in the study.
2. Clinical diagnosis of Amyotrophic Lateral Sclerosis (ALS).
3. Male or female patients between 18 to 80 years (inclusive).
4. Forced Vital Capacity (FVC) 65% of predicted value for gender, height and age at screening.
5. Evaluated with ALSFRS-R and Norris clinical rating scales for at least the past 4 weeks before study drug administration.

Exclusion criteria

1. Unable to understand information about the study or are expected not to collaborate with the study team.
2. Concurrent serious disease, other than ALS, at the discretion of the nvestigator.
3. Pregnancy.
4. Patients of childbearing potential not willing to use adequate double contraception with less than 1 percentage failure rate after the screening visit until the last visit.
5. Addiction to drugs or alcohol.
6. Confirmed HIV, hepatitis B or hepatitis C.
7. Known bleeding disorders or abnormal bleeding events.
8. Treatment with anticoagulant drugs warfarin and novel oral anticoagulants (NOAC) within the last 14 days prior to screening.
9. Treatment with Riluzole or Lamotrigine within the last 28 days prior to study drug administration.
10. Hypersensitivity to dextran sulfate.
11. Poor venous access.
12. Patients with clinically significant abnormal PK-INR, fibrinogen, von Willebrand factor and activated partial thromboplastin time (APTT) at screening.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2018-08-15 (Actual); Primary Completion 2019-08-20 (Actual); Study Completion 2019-08-20 (Actual)

PRIMARY OUTCOMES:
Frequency, seriousness and intensity of Treatment-emergent Adverse Events (TEAEs) | up to 3 months
  A TEAE is any adverse event (AE) not present prior to the initiation of IMP administration or any event already present that worsens in either intensity or frequency following exposure to the IMP. AEs (including baseline events) identified using any of the following methods will be recorded:
  * AEs spontaneously reported by the subject
  * AEs observed by the Investigator or medical personnel
  * AEs elicited based on non-leading questions from the Investigator or medical personnel
Change in physical status | up to 3 months
  A complete physical examination according to clinical praxis will be performed, including assessment of the head, eyes, ears, nose, throat (EENT), cardiac, peripheral vascular, pulmonary, musculoskeletal, neurologic, abdominal, lymphatic and dermatological functions.
  According to clinical praxis each function is judged as either normal or abnormal, and either clinically significant (CS) or not clinically significant (NCS)
  Change from baseline at 3 months.
Change in vital signs - blood pressure | up to 3 months
  Percent change in blood pressure (mmHg) from baseline at 3 months
Change in electrocardiogram (ECG) recordings | up to 3 months
  Change in single 12-lead ECG (PQ/PR (ms), QRS (ms), QT (ms) and QTcF (ms)) from baseline at 3 months
Change in vital signs - heart rate | up to 3 months
  Percent change in heart rate (bpm, beats per minute) from baseline at 3 months
Change in vital signs - body temperatue | up to 3 months
  Percent change in body temperature (degrees Celsius) from baseline at 3 months
Change in safety laboratory measurements - sodium, potassium, chloride, calcium, glucose (non-fasting) | up to 3 months
  According to clinical praxis, laboratory tests for sodium, potassium, chloride, calcium, glucose (non-fasting) will be analysed. Unit of measure is mmol/L
  According to clinical praxis each function is judged as either normal or abnormal, and either clinically significant (CS) or not clinically significant (NCS)
  Change from baseline at 3 months.
Change in safety laboratory measurements - albumin | up to 3 months
  According to clinical praxis, laboratory test for albumin will be analysed. Unit of measure is g/L
  According to clinical praxis each function is judged as either normal or abnormal, and either clinically significant (CS) or not clinically significant (NCS)
  Change from baseline at 3 months.
Change in safety laboratory measurements - AST, ALT, CK, alkaline phosphatase | up to 3 months
  According to clinical praxis, laboratory tests for aspartate amino-transferase (AST), alanine amino-transferase (ALT), creatine kinase (CK) and alkaline phosphatase will be analysed. Unit of measure is micro-kat/L
  According to clinical praxis each function is judged as either normal or abnormal, and either clinically significant (CS) or not clinically significant (NCS)
  Change from baseline at 3 months.
Change in safety laboratory measurements - creatinine and total bilirubin | up to 3 months
  According to clinical praxis, laboratory tests for creatinine and total bilirubin will be analysed. Unit of measure is micro-mol/L
  According to clinical praxis each function is judged as either normal or abnormal, and either clinically significant (CS) or not clinically significant (NCS)
  Change from baseline at 3 months.
Change in safety laboratory measurements - myoglobin | up to 3 months
  According to clinical praxis, laboratory test for myoglobin will be analysed. Unit of measure is micro-g/L
  According to clinical praxis each function is judged as either normal or abnormal, and either clinically significant (CS) or not clinically significant (NCS)
  Change from baseline at 3 months.
Change in safety laboratory measurements - CRP | up to 3 months
  According to clinical praxis, laboratory test for C-reactive protein (CRP) will be analysed. Unit of measure is milli-g/L
  According to clinical praxis each function is judged as either normal or abnormal, and either clinically significant (CS) or not clinically significant (NCS)
  Change from baseline at 3 months.
Change in hematology laboratory measurements - Hemoglobin and fibrinogen | up to 3 months
  According to clinical praxis, laboratory tests for hemoglobin (Hb) and fibrinogen will be analysed. Unit of measure is g/L
  According to clinical praxis each function is judged as either normal or abnormal, and either clinically significant (CS) or not clinically significant (NCS)
  Change from baseline at 3 months.
Change in hematology laboratory measurements - Red blood cell count | up to 3 months
  According to clinical praxis, laboratory test for blood cell count (RBC) will be analysed. Unit of measure is 10x12/L
  According to clinical praxis each function is judged as either normal or abnormal, and either clinically significant (CS) or not clinically significant (NCS)
  Change from baseline at 3 months.
Change in hematology laboratory measurements - WBC, platelets, basophils, eosinophils, lymphocytes, monocytes, neutrophils | up to 3 months
  According to clinical praxis, laboratory tests for white blood cell count (WBC), platelets, basophils, eosinophils, lymphocytes, monocytes and neutrophils will be analysed. Unit of measure is 10x9/L
  According to clinical praxis each function is judged as either normal or abnormal, and either clinically significant (CS) or not clinically significant (NCS)
  Change from baseline at 3 months.
Change in hematology laboratory measurements - APTT | up to 3 months
  According to clinical praxis, laboratory test for activated partial thromboplastin time (aPTT) will be analysed. Unit of measure is s
  According to clinical praxis each function is judged as either normal or abnormal, and either clinically significant (CS) or not clinically significant (NCS)
  Change from baseline at 3 months.
Change in hematology laboratory measurements - PK-INR | up to 3 months
  According to clinical praxis, laboratory test for prothrombin kinase international normalized ratio (PK-INR) will be analysed. Unitless measure
  According to clinical praxis each function is judged as either normal or abnormal, and either clinically significant (CS) or not clinically significant (NCS)
  Change from baseline at 3 months.

SECONDARY OUTCOMES:
Change in functional rating with Amyotrophic Lateral Sclerosis Functional Rating Scale - Revised (ALSFRS-R) | up to 3 months
  The ALSFRS-R provides a physician-generated estimate of the patient's degree of functional impairment, which can be evaluated serially to objectively assess any response to treatment or progression of disease. The ALSFRS-R includes questions that ask the physician to rate his/her impression of the patients level of functional impairment in performing one of twelve common tasks. Each task is rated on a five-point scale from 0 = can't do, to 4 = normal ability. Individual item scores are summed to produce a reported score of between 0=worst and 48=best
  Absolute change from baseline at 3 months
Change in functional rating with Norris rating scale | up to 3 months
  The Norris rating scale provides a physician-generated estimate of the patient's degree of functional impairment, which can be evaluated serially to objectively assess any response to treatment or progression of disease. The Norris rating scale includes questions that ask the physician to rate his/her impression of the patients level of functional impairment in performing one of 34 common tasks and bodily functions. Each task or function is rated on a four-point scale from 0 = can't do, to 3 = normal ability. Individual item scores are summed to produce a reported score of between 0=worst and 100=best
  Absolute change from baseline at 3 months
Change in pulmonary function (FVC) from baseline | up to 3 months
Change in Quality of Life (QoL) assessed by visual analogue scale (VAS) | up to 1.5 months
  Questionnaire with three questions for patient and next-of-kin self reporting of:
  * general health status
  * physical health status
  * mental health status
  Each item is rated on a millimeter scale from 0 = very bad, to 100 = very good
  Absolute change from baseline at 3 months
Change in functional rating of autonomous and sensory symptoms | up to 3 months
  The autonomous and sensory rating scale provides a physician-generated estimate of the patient's degree of functional impairment, which can be evaluated serially to objectively assess any response to treatment or progression of disease. The rating scale includes questions that ask the physician to rate his/her impression of the patients level of impairment in 16 autonomous and sensory functions. Each function is rated on a four-point scale from 0 = not impaired, to 3 = very impaired.
  Absolute change from baseline at 3 months
Change in maximum plasma concentration (Cmax) of ILB | up to 1 month
Change in exposure (Area Under the Curve, AUC) of ILB | up to 1 month
Changes in APTT (effect APTT) from day of dosing (day 1) | up to 1 month
Change in plasma concentration of hepatocyte growth factor (HGF) | up to 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, Sweden

REFERENCES:
- [Result] Logan A, Nagy Z, Barnes NM, Belli A, Di Pietro V, Tavazzi B, Lazzarino G, Lazzarino G, Bruce L, Persson LI. A phase II open label clinical study of the safety, tolerability and efficacy of ILB(R) for Amyotrophic Lateral Sclerosis. PLoS One. 2022 May 25;17(5):e0267183. doi: 10.1371/journal.pone.0267183. eCollection 2022. PMID 35613082
- [Result] Lazzarino G, Mangione R, Belli A, Di Pietro V, Nagy Z, Barnes NM, Bruce L, Ropero BM, Persson LI, Manca B, Saab MW, Amorini AM, Tavazzi B, Lazzarino G, Logan A. ILB(R) Attenuates Clinical Symptoms and Serum Biomarkers of Oxidative/Nitrosative Stress and Mitochondrial Dysfunction in Patients with Amyotrophic Lateral Sclerosis. J Pers Med. 2021 Aug 14;11(8):794. doi: 10.3390/jpm11080794. PMID 34442438